CLINICAL TRIAL: NCT00454740
Title: An Open-Label Multicenter Study to Assess the Efficacy and Safety of Daily Oral Administration of 5 and 10mg VESIcare® (Solifenacin Succinate) in Patients Who Wish to Switch From Detrol LA® (Tolterodine Tartrate Extended Release) for the Treatment of Overactive Bladder Symptoms Versus: VESIcare® Efficacy and Research Study US
Brief Title: Efficacy & Safety Study of VESIcare® (Solifenacin Succinate) in Patients Wishing to Switch From Detrol LA® for Treatment of Overactive Bladder
Acronym: VERSUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 905-UC-006
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Urinary Bladder, Overactive
Keywords: Urinary Bladder, Overactive; Urgency; VESIcare®; Solifenacin succinate
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: solifenacin succinate

INTERVENTIONS:
Drug: solifenacin succinate — Oral
  Other Names: VESIcare(R), YM905

SUMMARY:
To evaluate the efficacy of 5 and10mg solifenacin succinate in patients with urgency who have OAB syndrome (urgency, with or without urge incontinence, usually with frequency and nocturia) and wish to switch from tolterodine tartrate extended release to solifenacin succinate due to lack of sufficient improvement in urgency episodes

ELIGIBILITY:
Inclusion Criteria:

* Patients with OAB who have been treated with tolterodine tartrate extended release for at least 4 weeks immediately preceding entry into the study, and wish to switch to solifenacin succinate due to lack of sufficient improvement in urgency episodes.
* Previous non-drug treatment of OAB is allowed if it has been established at least 4 weeks prior to Screening and is continued throughout the study.
* At least 3 urinary urgency episodes/24 hours while receiving tolterodine tartrate extended release documented in a 3-day patient diary in the pre-washout assessments on tolterodine tartrate extended release with or without urge incontinence described as OAB syndrome.
* Prior to treatment with tolterodine tartrate extended release, patients must have had OAB syndrome for 3 or more months.

Exclusion Criteria:

* Previous treatment with darifenacin
* Treatment with tolterodine tartrate extended release for less than 4 weeks prior to enrollment in the study.
* Significant stress incontinence or mixed stress/urge incontinence where stress is the predominant factor as determined by the investigator.
* Evidence of a urinary tract infection; chronic inflammation such as interstitial cystitis and bladder stones.
* Clinically significant outflow obstruction as determined by the Investigator
* Uncontrolled narrow angle glaucoma, urinary or gastric retention.
* All patients with severe renal or hepatic impairment will be excluded
* Patients with chronic severe constipation or history of diagnosed gastrointestinal obstructive disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2004-06; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of 5 and 10mg solifenacin succinate in patients with urgency who have OAB syndrome. | Weeks 1, 4, 8 and 12

SECONDARY OUTCOMES:
To assess the improvement in urge incontinence, frequency,nocturia, and urgency | Weeks 1, 4, 8 and 12
Number of patients satisfied with treatment | Weeks 1, 4, 8 and 12
Assessment of efficacy | End of study
Evaluation of the safety and tolerability | Baseline to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (93):
- United States (93):
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - Dinuba, California
  - Glendora, California
  - La Mesa, California
  - Los Angeles, California
  - Mission Hills, California
  - Modesto, California
  - San Bernadino, California
  - Torrance, California
  - Upland, California
  - Valley Village, California
  - Aurora, Colorado
  - Denver, Colorado
  - Farmington, Connecticut
  - Norwalk, Connecticut
  - Trumbull, Connecticut
  - Waterbury, Connecticut
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Gainesville, Florida
  - Margate, Florida
  - New Port Richey, Florida
  - Orange City, Florida
  - Orlando, Florida
  - Saint Augustine, Florida
  - Tallahassee, Florida
  - Alpharetta, Georgia
  - Atlanta, Georgia
  - Blue Ridge, Georgia
  - Boise, Idaho
  - Coeur d'Alene, Idaho
  - Centralia, Illinois
  - Chicago, Illinois
  - Kankakee, Illinois
  - Niles, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Jeffersonville, Indiana
  - Muncie, Indiana
  - Baltimore, Maryland
  - Garrison, Maryland
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Edison, New Jersey
  - Lawrenceville, New Jersey
  - Neptune City, New Jersey
  - West Orange, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Bay Shore, New York
  - Brooklyn, New York
  - Garden City, New York
  - Lewiston, New York
  - New York, New York
  - Williamsville, New York
  - Cary, North Carolina
  - Concord, North Carolina
  - Hickory, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Bethany, Oklahoma
  - Tulsa, Oklahoma
  - Springfield, Oregon
  - Allentown, Pennsylvania
  - Bethlehem, Pennsylvania
  - Media, Pennsylvania
  - Monroeville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Aiken, South Carolina
  - Charleston, South Carolina
  - Myrtle Beach, South Carolina
  - Jefferson City, Tennessee
  - Arlington, Texas
  - Athens, Texas
  - Carrollton, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Bountiful, Utah
  - Layton, Utah
  - Ogden, Utah
  - Alexandria, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Spokane, Washington
  - Huntington, West Virginia
  - Madison, Wisconsin

REFERENCES:
- [Background] Chancellor MB, Zinner N, Whitmore K, Kobashi K, Snyder JA, Siami P, Karram M, Laramee C, Capo' JP Jr, Seifeldin R, Forero-Schwanhaeuser S, Nandy I. Efficacy of solifenacin in patients previously treated with tolterodine extended release 4 mg: results of a 12-week, multicenter, open-label, flexible-dose study. Clin Ther. 2008 Oct;30(10):1766-81. doi: 10.1016/j.clinthera.2008.10.011. PMID 19014833
- [Background] Zinner N, Noe L, Rasouliyan L, Marshall T, Seifeldin R. Impact of solifenacin on resource utilization, work productivity and health utility in overactive bladder patients switching from tolterodine ER. Curr Med Res Opin. 2008 Jun;24(6):1583-91. doi: 10.1185/03007990802081766. Epub 2008 Apr 17. PMID 18423103
- [Background] Swift SE, Siami P, Forero-Schwanhaeuser S. Diary and patient-reported outcomes in patients with severe overactive bladder switching from tolterodine extended release 4 mg/day to solifenacin treatment: An open-label, flexible-dosing, multicentre study. Clin Drug Investig. 2009;29(5):305-16. doi: 10.2165/00044011-200929050-00003. PMID 19366272
- [Background] Zinner N, Noe L, Rasouliyan L, Marshall T, Runken MC, Seifeldin R. Impact of solifenacin on quality of life, medical care use, work productivity, and health utility in the elderly: an exploratory subgroup analysis. Am J Geriatr Pharmacother. 2009 Dec;7(6):373-82. doi: 10.1016/j.amjopharm.2009.11.004. PMID 20129258
- [Derived] Capo' JP, Lucente V, Forero-Schwanhaeuser S, He W. Efficacy and tolerability of solifenacin in patients aged >/= 65 years with overactive bladder: post-hoc analysis of 2 open-label studies. Postgrad Med. 2011 Jan;123(1):94-104. doi: 10.3810/pgm.2011.01.2250. PMID 21293089